CLINICAL TRIAL: NCT07009834
Title: Solutions to the Challenges of Conduction System Pacing
Acronym: CSA
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 23HH8267
Record Dates: First submitted 2025-05-07; First posted 2025-06-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Conduction System Pacing; Pacing Therapy
Keywords: Challenges of conduction system pacing; CSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Derivation: These patients will undergo the research protocol. In these patients, the investigators will attempt to implant a permanent conduction system pacing lead, in lieu of the RV or LV lead. The lead will be implanted by operators who have implanted more than 40 leads to overcome the learning curve.
- Validation: These patients will undergo a conduction system pacemaker as standard clinical practice. The implanters will prospectively apply the step-by-step algorithm derived above to implant the conduction system lead using standard equipment alone; fluoroscopy, PSA and 12-lead ECG. The investigators will assess the success rate, conduction system capture threshold, procedure time and fluoroscopy time. Although all operators will be highly experienced device implanters, these implants will include operators who are new to conduction system lead implantation.
- 2-lead ECG group: Patients with a chronic conduction system lead implant under device follow-up will under go 2-lead ECG of multiple pacing and sensing configurations. These patients will be attending for routine appointments. The pacing and sensing configurations are undertaken as part of routine checks.

SUMMARY:
Conduction system pacing is a new way of stimulating the heart using pacemaker wires. Traditional pacemakers stimulate the heart muscle which causes disordered heart beats: the walls of the heart move at different times. This wears down the heart over time.

Conduction system pacemakers stimulate the heart's electrical system directly producing natural heart beats that are much less disordered. Unfortunately, these pacemakers can only be implanted by a small group of experts at specialised centres with specialist equipment. This study aims to allow conduction system pacemakers to be offered to any patient at any hospital by simplifying the process of inserting the pacemaker wires and the improving the pacemaker's ability to interpret electrical traces.

Firstly, the best locations in the heart for conduction system pacemaker wires using specialised electrical traces, MRI and ultrasound scans will be identified. Features that can be seen on X-ray to guide doctors to these locations will then be identified. Secondly, the investigators will collect electrical information from the pacemaker wires and additional electrical traces to develop an algorithm that can make the interpretation the electrical traces more accurate.

DETAILED DESCRIPTION:
Study A:

100 patients will be prospectively recruited. These patients will be further divided into a derivation and validation group. The derivation group will consist of the first fifty patients recruited (patients 1-50) and the validation group will consist the second fifty patients recruited (patients 51-100).

All 100 patients will have an indication for pacemaker insertion and will undergo a conduction system pacemaker implant.

The derivation group will undergo the research protocol which will include additional measurements from:

1. Ultra-high frequency ECG. A non-invasive surface ECG that detects, isolates and amplifies high frequency components that are filtered out in conventional ECGs.
2. Electro-anatomical mapping. In majority of participants, the invasive mapping catheter will be inserted from the same venous access point to collect detailed electrical and anatomical data. In a small subset of patients, activation maps of the left ventricle will be collected, where the access will be through the femoral artery in the groin.

   Non invasive mapping will also be performed in a subgroup of patients with ECGi, where the participants will wear a 252 electrode ECG vest during the procedure. These patients will undergo a pre-procedural CT scan with the vest.
3. Echocardiography. Participants will undergo either transthoracic echocardiography, transoesophageal echocardiography or intracardiac echocardiography.

   Additional venous access from the femoral vein in the groin will be sought for patients undergoing intracardiac echocardiography.
4. Haemodynamic assessment Invasive blood pressure will be obtained in patients who already have arterial access for the left ventricular electro- anatomical maps. The sheath will be connected to the pressure inducer. Non invasive beat-by-beat blood pressure will be obtained by a high precision finger cuff (finometer).

A further 50 patients will be prospectively recruited that will make up the validation cohort for Study A. These patients will undergo a conduction system pacemaker as standard clinical practice. The step-by-step algorithm will be prospectively derived from the above to implant the conduction system lead using standard equipment alone; fluoroscopy, PSA and 12-lead ECG. The success rate, conduction system capture threshold, procedure time and fluoroscopy time will be assessed. Although all operators will be highly experienced device implanters, these implants will include operators who are new to conduction system lead implantation.

Study B:

In patients 1-50 undergoing implantation of conduction system pacemakers, 2-lead surface ECG alongside conventional lead data will be collected. A surface 12-lead ECG will be collected as well. The patients will undergo the standard pacing manoeuvres for conduction system pacing. The patient will be paced using the PSA and a 12-lead ECG and 2-lead ECG will be collected via Bard, a computer software that is able to collect highly accurate ECG traces of the heart using mapping catheters placed inside the heart and the surface ECG.

Prospective data from 200 patients with a chronic conduction system lead implant under device follow-up to obtain EGM, 12 -lead ECG and the 2-lead ECG recordings of multiple pacing and sensing configurations will also be collected. These patients will be attending for routine appointments. The pacing and sensing configurations are undertaken as part of routine checks

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a ventricular pacing indication: high grade atrioventricular block and symptomatic trifasicular, bifasicular block or left bundle branch block LBBB for cardiac resynchronisation therapy
2. Adults willing to take part (ages 18 - 100 years old)
3. Able to give consent.

Exclusion Criteria:

1. Unable to give consent
2. Children age < 18 years and adults > 100 years old
3. Pregnant patients As per standard of care, female patients of child-bearing age will have a urine pregnancy test prior to their procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from London who are attending Hammermsith Hospital for device therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
A1: Success rates of conduction system lead implant (novel workflow vs conventional methods) | From enrollment until 6 months after recruitment of last patient
B1: The number of patients with morphology change seen during decrementing output threshold test of 2-lead ECG when compared to gold standard 12-lead ECG | From enrollment until 6 months after recruitment of last patient

SECONDARY OUTCOMES:
A2: Procedure and fluoroscopy times of the streamlined workflow to current conventional methods of His-bundle and Left-bundle pacing | From enrolment to until completion of PPM insertion of the last patient recruited into Study A (patient 100); average total of 3 years
A2: Procedure and fluoroscopy times of the streamlined workflow of conduction system implant to current right ventricular pacing | From enrolment to until completion of PPM insertion of the last patient recruited into Study A (patient 100); average total of 3 years
A2: Assess capture threshold of conduction system pacing from the optimised workflow to that of conventional methods of conduction system implantation | From enrollment until 6 months after recruitment of last patient
  Threshold is measured through the device, looking to achieve the minimum energy (in V) required to safely and reliably capture the cardiac tissue target. In this outcome, the investigators will compare the minimum threshold required to achieve capture of conduction system pacing to that of conventional right ventricular pacing and asses if this the same, higher or lower.
A2: Define left bundle area capture diagnostics and delineate differences between left ventricular septal pacing. | From enrollment until 6 months after recruitment of last patient
B2: Improvement in device battery life measured in days and months with novel device algorithm applied | From enrollment until 6 months after recruitment of last patient
  Device battery time is given upon device interrogation and is dependent on percentage of the time the patient is paced and the energy delivered. Battery life will increase if less energy is required. The investigators will assess if there is a increase in days or months in the battery life of the pacemaker with introduction of the novel algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Whinnett, BM.BS, Principal Investigator — Imperial College London, Imperial College Healthcare Trust
Locations (1):
- Imperial College Healthcare Trust; Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT07009834/Prot_000.pdf